CLINICAL TRIAL: NCT00915590
Title: Topical IL-1-Ra for Treatment of Corneal Neovascularization
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Reza Dana, MD (Other)
Responsible Party: Sponsor-Investigator, Reza Dana, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-03-017; Protocol #09-03-017 (Other: Massachusetts Eye and Ear Infirmary)
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo first, then IL-1RA (Experimental): It is our intent that 10 patients will complete a course of treatment with placebo, followed by a course of treatment with 5% custom made topical IL-1Ra.
  Interventions: Drug: Placebo; Drug: IL-1Ra
- IL-1RA first, then Placebo (Experimental): It is our intent that 10 patients will complete a course of treatment with 5% custom made topical IL-1Ra, followed by a course of treatment with placebo
  Interventions: Drug: Placebo; Drug: IL-1Ra

INTERVENTIONS:
Drug: Placebo — Custom eye drop eye three times a day in both eyes for a period of 6 weeks
Drug: IL-1Ra — 5% custom made topical IL-1Ra 3 times a day in both eyes for a period of 6 weeks
  Other Names: Kineret

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of Interleukin-1-Receptor Antagonist eye drops for the treatment of corneal blood vessels.

DETAILED DESCRIPTION:
Normally avascular, under many pathologic conditions, vessels may invade the cornea from the limbal vascular plexus. Infection, inflammation, ischemia, degeneration, or trauma, and the loss of the limbal stem cell barrier can cause corneal neovascularization. Growth of new vessels may result in corneal scarring, edema, lipid deposition, and inflammation that may alter visual acuity and is a leading cause of monocular visual impairment and blindness. Additionally, it results in the loss of immune response across the cornea, thereby worsening the prognosis of a subsequent penetrating keratoplasty (PK). Growth of new blood and lymphatic vessels from preexisting vessels are mediated by members of the vascular endothelial growth factor (VEGF) family. This study is designed to investigate whether Interleukin-1-Receptor Antagonist is a drug that is both safe and effective in blocking VEGF pathways, stopping new growth, and reducing old vessel growth.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Patients with superficial or deep corneal NV that extends farther than 1 mm from the limbus
* Patients are in generally good stable overall healthExclusion Criteria: • Has received treatment with anti-VEGF agents (topical, intraocular or systemic) within 30 days of study entry
* Corneal or ocular surface infection within 30 days prior to study entry• Ocular or periocular malignancy
* Contact lens (excluding bandage contact lens) use within 2 weeks prior to study entry
* Persistent epithelial defect (>1mm and ≥14 days duration) within 2 weeks prior to study entry
* Intravitreal or periocular steroids within 2 weeks prior to study entry
* Change in dose/frequency of topical steroids and/or NSAIDs within 2 weeks prior to study entry
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using contraception
* Signs of current infection, including fever and current treatment with antibiotics
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, MD, MPH, MSc, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in this study were recruited from Mass. Eye and Ear Infirmary from May 2009 - February 2010.
Pre-assignment Details: This is a single site, randomized, double masked, crossover, phase I/II study of topical IL-1Ra (5.0%) in subjects with corneal neovascularization.
Groups:
- Placebo First, Then IL-1Ra: 10 patients will complete a course of treatment with placebo, followed by a course of treatment with 5% custom made topical IL-1Ra.
  IL-1Ra : 5% custom made topical IL-1Ra 3 times a day in both eyes for a period of 6 weeks
  Placebo : Custom eye drop eye three times a day in both eyes for a period of 6 weeks
- IL-1Ra First, Then Placebo: 10 patients will complete a course of treatment with 5% custom made topical IL-1Ra, followed by a course of treatment with placebo
  IL-1Ra : 5% custom made topical IL-1Ra 3 times a day in both eyes for a period of 6 weeks
  Placebo : Custom eye drop eye three times a day in both eyes for a period of 6 weeks
Period: Overall Study
Arm/Group | Placebo First, Then IL-1Ra | IL-1Ra First, Then Placebo
Started | 5 | 5
Completed | 3 | 4
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then IL-1Ra | IL-1Ra First, Then Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (24) | 66 (19) | 56 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular Adverse Event
Description: Incidence and severity of ocular adverse events, as identified by eye examination and visual acuity testing.
Time Frame: 64 Weeks
Measure: Number; unit: participants
Groups:
- Placebo First, Then IL-1RA: It is our intent that 10 patients will complete a course of treatment with placebo, followed by a course of treatment with 5% custom made topical IL-1Ra.
  IL-1Ra : 5% custom made topical IL-1Ra 3 times a day in both eyes for a period of 6 weeks
  Placebo : Custom eye drop eye three times a day in both eyes for a period of 6 weeks
- IL-1RA First, Then Placebo: It is our intent that 10 patients will complete a course of treatment with 5% custom made topical IL-1Ra, followed by a course of treatment with placebo
  IL-1Ra : 5% custom made topical IL-1Ra 3 times a day in both eyes for a period of 6 weeks
  Placebo : Custom eye drop eye three times a day in both eyes for a period of 6 weeks
Arm/Group | Placebo First, Then IL-1RA | IL-1RA First, Then Placebo
Number analyzed (Participants) | 5 | 5
participants | 2 | 3

2. Primary Outcome: Extent of Neovascular Area (NA)
Description: The Principal Investigator decided to terminate the study and stop enrollment because of difficulty recruiting subjects. Although data were collected for this Outcome Measure, no analysis was performed. All records were destroyed following the required retention period. Data are no longer available for analysis.
Time Frame: 64 weeks
Population: The Principal Investigator decided to terminate the study and stop enrollment because of difficulty recruiting subjects. Although data were collected for this Outcome Measure, no analysis was performed. All records were destroyed following the required retention period. Data are no longer available for analysis.
Arm/Group | Placebo First, Then IL-1RA | IL-1RA First, Then Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Vessel Caliber (VC), Measuring the Mean Diameter of the Corneal Vessels
Description: as for outcome 2
Time Frame: 64 Weeks
Population: as for outcome 2
Arm/Group | Placebo First, Then IL-1Ra | IL-1Ra First, Then Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Invasion Area (IA), Measuring the Fraction of the Total Corneal Area Invaded by the Vessels
Description: as for outcome 2
Time Frame: 64 Weeks
Population: as for outcome 2
Arm/Group | Placebo First, Then IL-1Ra | IL-1Ra First, Then Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Best Spectacle-Corrected Visual Acuity (BSCVA)
Description: as for outcome 2
Time Frame: 64 weeks
Population: as for outcome 2
Arm/Group | Placebo First, Then IL-1Ra | IL-1Ra First, Then Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Central Corneal Thickness
Description: as for outcome 2
Time Frame: 64 Weeks
Population: as for outcome 2
Arm/Group | Placebo First, Then IL-1Ra | IL-1Ra First, Then Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 9 month period (May 2009 - February 2010).
Groups:
- Placebo: Placebo : Custom eye drop eye three times a day in both eyes for a period of 6 weeks
- IL-1Ra: IL-1Ra : 5% custom made topical IL-1Ra 3 times a day in both eyes for a period of 6 weeks
- Off Treatment: Off treatment
Arm/Group | Placebo | IL-1Ra | Off Treatment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 1/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | IL-1Ra (N=10) | Off Treatment (N=10)
Itchy Eyes (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Eye Redness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diminished Vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular Herpes Flare-up (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gall Bladder Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment goal for this study was set at 20 participants (10 for each treatment arm). After an interim analysis, the Principal Investigator decided to terminate the study and stop enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No